CLINICAL TRIAL: NCT00676325
Title: A Randomized Controlled Trial Study, To Compare Colporrhaphy Versus NAZCA TC™ ,Macroporous Polypropylene Mesh, In Surgical Treatment To Greater Anterior Vaginal Prolapse .
Brief Title: Surgical Treatment To Greater Anterior Vaginal Prolapse
Acronym: Nazcatc™
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of São Paulo (Other)
Responsible Party: carlos antonio del roy, federal university of sao paulo- unifesp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: unifespcep 1790/06
Record Dates: First submitted 2008-05-01; First posted 2008-05-13 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Hernia; Cystocele
Keywords: anterior vaginal prolapse; traditional treatment; mesh, graft; NAZCA TC™ POP REPAIR SYSTEM; colporrhaphy
MeSH Terms: conditions — Hernia; Cystocele | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Women 50 years and older with greater anterior vaginal prolapse,whit stress incontinence or not, requiring surgical correction were eligible for participation.traditional colporrhaphy in this group.
  Interventions: Procedure: Surgical treatment of Anterior Vaginal Prolapse; Device: NAZCA TC™ POP REPAIR SYSTEM ,promedon® , argentina.
- 2 (Active Comparator): The NAZCA TC™ POP REPAIR SYSTEM (polypropylene mesh repair),promedon™ , cordoba, argentina, is used to repair anterior vaginal prolapse by a transobturator and pre pubic approach . Helical needles are used to anchor graft to the pelvic sidewall at two points transobturator, the other two arms pre pubic needles is used. We designed this randomized control trial to compare the anatomic success rates, effect on quality of life and sexual symptom scores, and rates of adverse events of the procedure with polypropylene mesh with that of anterior colporrhaphy, with planned follow-up of 1 years.
  Interventions: Procedure: Surgical treatment of Anterior Vaginal Prolapse; Device: NAZCA TC™ POP REPAIR SYSTEM ,promedon® , argentina.; Procedure: surgical treatment for anterior vaginal wall prolapse

INTERVENTIONS:
Procedure: Surgical treatment of Anterior Vaginal Prolapse — seventy patients with greater anterior vaginal prolapse, whit stress incontinence or not, were randomly assigned to either colporrhaphy or polypropylene mesh repair (NAZCA TC™ POP REPAIR SYSTEM ) . The primary outcome was recurrent anterior vaginal prolapse, and secondary outcomes were effects on quality of life and sexual symptom scores, operative time, blood loss, length of hospitalization, and adverse events.
  Other Names: traditional colporraphy anterior vaginal wall; polypropylene mesh - NAZCA TC™ POP REPAIR SYSTEM
Device: NAZCA TC™ POP REPAIR SYSTEM ,promedon® , argentina. — Women 50 years and older with greater anterior vaginal prolapse,whit stress incontinence or not, requiring surgical correction .
  Other Names: traditional colporraphy
Procedure: surgical treatment for anterior vaginal wall prolapse — Women 50 years and older with greater anterior vaginal prolapse,whit stress incontinence or not requiring surgical correction were eligible for participation.
  Other Names: NAZCA TC™ POP REPAIR SYSTEM
  Arms: 2

SUMMARY:
A RCT study to compare traditional colporrhaphy versus polypropylene mesh in treatment of the anterior vaginal wall prolapse.

DETAILED DESCRIPTION:
Seventy patients with greater anterior vaginal prolapse, whit stress incontinence or not, were randomly assigned to either colporrhaphy or polypropylene mesh repair( NAZCA TC™ POP REPAIR SYSTEM) . The primary outcome was recurrent anterior vaginal prolapse, and secondary outcomes were effects on quality of life and sexual symptom scores, operative time, length of hospitalization, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Women 50 years and older with greater anterior vaginal prolapse,whit stress incontinence or not,point (Ba)ics96, below hymenal ring requiring surgical correction were eligible for participation.

Exclusion Criteria:

Patients were excluded if they had:

* Stage 0 or I (ics96) anterior vaginal support
* Declined participation
* Were pregnant or contemplating future pregnancy
* Had prior anterior vaginal prolapse repair with biologic or synthetic graft
* Active or latent systemic infection
* Compromised immune system
* Uncontrolled diabetes mellitus,
* Previous pelvic irradiation or cancer
* Known hypersensitivity to polypropylene.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is recurrent anterior vaginal prolapse | 1 year

SECONDARY OUTCOMES:
Secondary outcomes are, first, operative time (from first incision to closure of last incision), blood loss (preoperative minus postoperative day one hemoglobin), length of hospitalization, adverse events, PQol , FSFI and Dyspareunia . | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: carlos a del roy, M D, Principal Investigator — Federal University of São Paulo
Locations (1):
- Sao Paulo Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Riccetto C, Miyaoka R, de Fraga R, Barbosa R, Dambros M, Teixeira A, Palma P. Impact of the structure of polypropylene meshes in local tissue reaction: in vivo stereological study. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Aug;19(8):1117-23. doi: 10.1007/s00192-008-0582-2. Epub 2008 Mar 20. PMID 18351281
- See also: INTERNATIONAL UROGYNECOLOGICAL ASSOCIATION — http://www.iuga.org